CLINICAL TRIAL: NCT05442437
Title: Clinical Study of Human Umbilical Cord Mesenchymal Stem Cells for Treating Decompensated Liver Cirrhosis Associated With HBV
Brief Title: Clinical Study of hUC-MSCs Treating Decompensated Liver Cirrhosis With HBV
Acronym: CS-hUC-MSCs
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 03
Record Dates: First submitted 2022-04-13; First posted 2022-07-05 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2021-12

CONDITIONS: HBV

STUDY DESIGN:
Intervention Model Description: We allocate 24 participants into 3 group, low-dose, medium-dose and high-dose group. It is going to proceeded sequential from low-dose group to high-dose group. Next group is allowed to be started only the last group has been finished.
  1. Low-dose group: 100mL human umbilical cord mesenchymal stem cell preparation, containing 2.5×10^7 cells;
  2. medium-dose group: 100mL human umbilical cord mesenchymal stem cell preparation, containing 5.0×10^7 cells;
  3. High-dose group: 100mL human umbilical cord mesenchymal stem cell preparation, containing 1.0×10^8 cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose group (Experimental): 100mL human umbilical cord mesenchymal stem cell preparation, containing 2.5×10^7 cells.
  Interventions: Biological: hUCMSCs
- medium-dose group (Experimental): 100mL human umbilical cord mesenchymal stem cell preparation, containing 5.0×10^7 cells.
  Interventions: Biological: hUCMSCs
- High-dose group (Experimental): 100mL human umbilical cord mesenchymal stem cell preparation, containing 1.0×10^8 cells.
  Interventions: Biological: hUCMSCs

INTERVENTIONS:
Biological: hUCMSCs — Human umbilical cord mesenchymal stem cell preparation, 100ml/ bag, containing 2.5×107 cells, 5.0×107 cells, 1.0 x 108 cells

SUMMARY:
The purpose of this study was to observe the safety ,tolerability ,Efficacy dose of human umbilical cord mesenchymal stem cells in patients of decompensated liver cirrhosis with HBV.

DETAILED DESCRIPTION:
Investigators plan to recruit 24 voluntary patients of decompensate liver cirrhosis with HBV, dividing them into 3 group：1) low-dose group: 100mL with 2.5×10^7 cells；2) medium-dose group: 100mL with 5.0×10^7 cells；3) high-dose group: 100mL with 1.0×10^8 cells. Each group contains 8 patients. Investigators treat the participants with human umbilical cord mesenchymal stem cells via venous transfusion. First investigators arrange a whole test for participants, such as vital sign examination, laboratory test, ECG, CT, MRI, ultrasound etc. Investigators screen these patients with a complete eligibility criteria. Then investigators proceed the therapy in the 1st, 8th and 15th day. There are 8 times of follow-up visit for these patients, 4 times of those are proceeded during the hospitalization, while other 4 times happens after the discharge. The follow-up visit includes vital sign examination, laboratory test, ECG, CT, MRI, ultrasound, Child-Pugh grade, MELD grade, SF-36 test. These follow-up visit last 24 weeks since the first treatment. After that, investigators also arrange a survival visit through phone or clinic each 6 months, lasting another 1.5 years. The main object of this research is investigating the survival rate, promotion of the liver function, improvement of health, safety of hUC-MSCs, tolerability of patients, for exploring a new way for the therapy of decompensated liver cirrhosis with HBV.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 (including 18 and 65), regardless of gender;
* Decompensated stage of viral hepatitis B cirrhosis;
* The effect of conventional medical treatment is not good, and the condition is repeated;
* ALB < 35g/L, TBIL < 170μmol/L, INR > 30%, Child-pugh score ≥7; MELD score ≤15;
* Hgb > 70g/L, PLT > 3×109/L;
* Unconditional acceptance for liver transplantation; 7）Participate in the clinical study voluntarily, cooperate with doctors to carry out the study, and sign informed consent.

Exclusion Criteria:

* With spontaneous peritonitis or other serious infection;
* Patients with hepatorenal syndrome;
* Severe hepatic encephalopathy, massive hemorrhage of digestive tract or varicose 4. vein in recent 1 month;
* Portal vein thrombosis; Complicated with serious diseases of heart, lung, kidney,
* blood and endocrine system;
* HIV positive;
* Positive autoantibodies related to autoimmune liver disease;
* Presence of liver or any type of malignant tumor;
* Pregnant women, breast-feeding women or those with recent birth plans;
* Those who have a history of alcohol and drug abuse and failed to get rid of it effectively;
* Participated in other clinical trials within 3 months prior to enrollment;
* Participated in clinical research on stem cells;
* Unwillingness to sign informed consent;
* Other conditions that the investigator considers inappropriate for patients to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Serum albumin in g/L | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
alanine aminotransferase in U/L | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
aspartate aminotransferase in U/L | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
cholinesterase in U/L | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Total bilirubin in μmol/L | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Direct bilirubin in μmol/L | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Serum cholesterol in mmol/L | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Prothrombin activity in percentage | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Antithrombin in mg/L | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.

SECONDARY OUTCOMES:
survival rate | 2 years
  survival rate after 2 years since the first therapy
Child-Pugh grade | 24 weeks
  Child-Pugh grade is defined according to hepatic encephalopathy, ascites，serum albumin, total bilirubin, prothrombin time. Score 5-6 is grade A. Score 7-9 is grade B. Score 10-15 is grade C.
  We compare the Child-Pugh grade in first day, 4th, 8th, 12th and 24th week, to describe its tendency.
Rate of weight change | 24 weeks
  We compare the weight in first day, 4th, 8th, 12th and 24th week, to describe its tendency.
Ascites | 24 weeks
  We test the ascites via ultrasound, CT and MRI. We classify the ascite level into none, low and high.
  We compare the Child-Pugh grade in first day, 4th, 8th, 12th and 24th week, to describe its tendency.
clinical symptoms | 24 weeks
  Including lower limb edema, hematemesis, jaundice, fatigue, poor appetite. We compare these symptoms in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Th1 cells in percentage | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Th2 cells in percentage | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Natural killer T cells in percentage | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Interleukin-1β cells in pg/mL | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Interleukin-4 cells in pg/mL | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Interleukin-6 cells in pg/mL | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Interleukin-8 cells in pg/mL | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Interleukin-12 cells in pg/mL | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Interleukin-15 cells in pg/mL | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Interleukin-17A cells in pg/mL | 24 weeks
  We compare this index in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Medical images | 24 weeks
  Ultrasound in first day, 4th, 8th, 12th and 24th; enhanced CT scanning and/or MRI-Primovist scanning in first day, 12th week and 24th week.
The Medical outcomes study 36-item Short Form Health Survay scale (SF-36 scale) | 24 weeks
  SF-36 scale is a measurement for patients' living quality. The scores contain 8 parts, including physical functioning, role-physica, bodily pain, general health, vitality, social functioning, role-emotional and mental health. Conversion score=(actual score-minimum score in this part)/(maximum score in this part-minimum score in this part)*100. Score of each part range from 0 to 100. The higher score means more healthy. We proceed SF-36 test in 12th week and 24th week
MELD score | 24 weeks
  MELD=3.78*Ln(total bilirubin mg/dL)+11.2*Ln(INR)+9.57*Ln(serum creatine mg/dL)+6.43 (for HBV patient) We compare MELD score in first day, 4th, 8th, 12th and 24th week, to describe its tendency.

OTHER OUTCOMES:
Adverse events | 24 weeks
  Including infusion reaction, anaphylaxis, hemolysis, acute liver failure, acute kidney failure. We observe whether participants shows these adverse event during the first whole 2 weeks and 4th, 8th, 12th and 24th weeks
Vital signs | 24 weeks
  body temperature, pulse, respiration, blood pressure. We measure the vital signs in first day, 1st , 2nd, 3rd, 4th, 8th, 12th and 24th week.
Physical examination | 24 weeks
  Including jaundice in skin or sclera, liver palms, spider angioma, abdominal tenderness, borborygms, shifting dullness. We proceed the physical examination in first day, 1st , 2nd, 3rd, 4th, 8th, 12th and 24th week.
Leukocyte in 10^9/L | 24 weeks
  We test it in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Hemoglobin in g/L | 24 weeks
  We test it in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Thrombocyte in 10^9/L | 24 weeks
  We test it in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Serum creatine in | 24 weeks
  We test it in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Serum creatine in μmol/L | 24 weeks
  We test it in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Serum urea nitrogen in mmol/L | 24 weeks
  We test it in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Alpha-fetoprotein in ng/mL | 24 weeks
  We test it in first day, 4th, 8th, 12th and 24th week, to describe their tendency.
Electrocardiogram of 12 leads | 24 weeks
  Including lead I, II, III, AVL, AVF, AVR, V1 to V6. We record the diagnosis of the ECG, not a specific parameter. We test it in first day, 4th, 8th, 12th and 24th week.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China